CLINICAL TRIAL: NCT06768853
Title: Clinical Study on Predicting Mediastinal Lymph Node Metastasis in Patients with Lung Cancer by the Predictive Model Based on Clinical Characteristics and Radiomics
Brief Title: The Accuracy of Targeted Lymph Node Dissection of Non-small Cell Lung Cancer Patients According to Predictive Models
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 20240329
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; mediastinal lymph node
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Model group (Experimental): During surgery, lymph nodes predicted to be metastatic will be dissected based on the predicted results of the model.
  Interventions: Procedure: Lymph node dissection based on the model
- Guideline group (Active Comparator): During surgery, lymph nodes will be dissected based on the NCCN guidelines (2023).
  Interventions: Procedure: Lymph node dissection based on the guidelines

INTERVENTIONS:
Procedure: Lymph node dissection based on the guidelines — During surgery, mediastinal lymph nodes will be dissected based on the NCCN guidelines (2023) .
  Arms: Guideline group
Procedure: Lymph node dissection based on the model — During surgery, lymph nodes will be dissected based on the predicted lymph node status by the model.
  Arms: Model group

SUMMARY:
Investigators combined the clinical and radiomics characteristics of resectable non-small cell lung cancer patients to construct an accurate model for preoperative prediction of mediastinal lymph node status. For the patients in the experimental group, lymph nodes will be dissected based on the predicted lymph node status by the model, while in the control group, the lymph nodes will be dissected according to the NCCN guidelines (2023). Investigators expect that performing lymph node dissection according to the predictive model can lead to better prognosis for patients.

DETAILED DESCRIPTION:
Investigators combined the clinical and radiomics characteristics of resectable non-small cell lung cancer patients to construct an accurate model for preoperative prediction of mediastinal lymph node status. Investigators will randomly divide all enrolled patients into an experimental group and a control group. For the patients in the experimental group, lymph nodes will be dissected based on the predicted lymph node status by the model, while in the control group, the lymph nodes will be dissected according to the NCCN guidelines (2023). Investigators will calculate the consistency between preoperative prediction results and postoperative pathological results to verify the accuracy of the model. And investigators will evaluate the impact of this new lymph node dissection method on prognosis by comparing the intraoperative blood loss, postoperative complications, disease-free survival, and overall survival between the two groups of patients. Investigators expect that performing lymph node dissection according to the predictive model can lead to better prognosis for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 70 years old;
2. Chest CT shows a single pulmonary nodule, which may be adenocarcinoma or squamous cell carcinoma;
3. Chest CT shows multiple pulmonary nodules, but preoperative evaluation suggests that pulmonary nodules other than the main lesion are benign;
4. Preoperative auxiliary examination evaluates the patient as clinically resectable lung adenocarcinoma or squamous cell carcinoma in stages I, II, or IIIA (UICC-TNM 9th edition);
5. ECOG score 0-1;
6. Preoperative lung function FEV1 ≥ 1.0L and actual/expected value ≥ 80%;
7. No contraindications for surgery;
8. Technically, lobectomy or segmental resection combined with lymph node dissection can be performed;
9. Preoperative plain scan and enhanced chest CT examination;
10. The interval between surgery and chest CT, lung function, and electrocardiogram examinations is less than or equal to 28 days;
11. The patient signs a written informed consent form.

Exclusion Criteria:

1. Chest CT suggests multiple primary lung cancer or metastatic cancer;
2. Previous history of thoracic surgery;
3. Previous history of malignant tumors;
4. History of neoadjuvant therapy;
5. A history of severe heart failure, myocardial infarction, cerebral infarction, and pneumonia within 6 months prior to surgery;
6. Concurrent active bacterial or fungal infections;
7. Severe underlying lung diseases such as interstitial lung disease, pulmonary fibrosis, or emphysema are complicated;
8. Concomitant mental illness;
9. Pregnant/lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Consistency rate between preoperative prediction results and postoperative pathological results | 1 week after surgery
  Compare postoperative lymph node pathology results with preoperative prediction results

SECONDARY OUTCOMES:
Postoperative complications | 30 days after surgery
  Observation of complications within 30 days after surgery
Postoperative recurrence rate | 2 years after surgery
  Observe for recurrence within 2 years after surgery
Disease-free survival | 2 years after surgery
  Follow up after surgery to determine if there is any recurrence or metastasis, and calculate disease-free survival
Overall survival | 2 years after surgery
  Follow up after surgery to determine if there is death, and calculate overall survival
Intraoperative blood loss | During the surgery
  Record intraoperative blood loss
Postoperative drainage volume | 2 weeks after surgery
  Record postoperative drainage volume
Postoperative drainage time | 2 weeks after surgery
  Record the time from the end of the surgery to the removal of the drain tube

CONTACTS AND LOCATIONS:
Overall Officials: Hexiao Tang, PhD, Study Chair — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No